CLINICAL TRIAL: NCT00419094
Title: A Multi-center, Double-blind, Historical Control, Randomized Conversion to Monotherapy Study With Keppra XR for Treatment of Partial Onset Seizures
Brief Title: Conversion to Monotherapy Study With Keppra XR for Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01280; 2007-000897-21 (EudraCT Number)
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy
Keywords: Keppra XR; conversion to monotherapy; partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keppra XR 1000 mg/day (Experimental): 1000 mg/day once daily for 18 weeks (administered as two levetiracetam XR tablets and two placebo tablets once daily)
  Interventions: Drug: Keppra XR
- Keppra XR 2000 mg/day (Experimental): 2000 mg/day once daily for 18 weeks (administered as four levetiracetam XR tablets once daily)
  Interventions: Drug: Keppra XR

INTERVENTIONS:
Drug: Keppra XR — Administered as two 500 mg tablets (1000 mg) and two placebo tablets once daily for 18 weeks
  Arms: Keppra XR 1000 mg/day
Drug: Keppra XR — Administered as four 500 mg tablets (2000 mg) once daily for 18 weeks
  Arms: Keppra XR 2000 mg/day

SUMMARY:
The primary objective of this study is to assess the efficacy of two doses of Keppra XR compared with a historical control as the placebo, in the monotherapy treatment of partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 12 to 75 years of age.
* Subjects must have inadequately controlled partial onset epilepsy.
* Subjects must be experiencing 2 to 40 seizures per 4-week period while being maintained on one or two standard AED(s)

Exclusion Criteria:

* A history of status epilepticus in the 6 months preceding randomization.
* Significant medical, psychiatric or neurological illness.
* Intake of benzodiazepines on more than an occasional basis
* History of previous treatment with levetiracetam or sensitivity to levetiracetam.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (45):
- United States (24):
  - Dothan, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Jacksonville, Florida
  - Loxahatchee Groves, Florida
  - Atlanta, Georgia
  - Suwanee, Georgia
  - Winfield, Illinois
  - Witchita, Kansas
  - Shreveport, Louisiana
  - Bethesda, Maryland
  - Detroit, Michigan
  - Camden, New Jersey
  - New Brunswick, New Jersey
  - Buffalo, New York
  - Cedarhurst, New York
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Monaca, Pennsylvania
  - Philadelphia, Pennsylvania
  - Beaufort, South Carolina
- Mexico (7):
  - Monterrey, Nuevo León
  - Aguascalientes
  - Distrio Federal
  - Guadalajara
  - Guadalajara Jalisco
  - Mexico City
  - Monterrey
- Poland (8):
  - Bialystok
  - Gdansk
  - Katowice
  - Lodz
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
- Russia (6):
  - Kalingrad
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara
  - Yaroslavl

REFERENCES:
- [Derived] Chung S, Ceja H, Gawlowicz J, Avakyan G, McShea C, Schiemann J, Lu S. Levetiracetam extended release conversion to monotherapy for the treatment of patients with partial-onset seizures: a double-blind, randomised, multicentre, historical control study. Epilepsy Res. 2012 Aug;101(1-2):92-102. doi: 10.1016/j.eplepsyres.2012.03.007. Epub 2012 Apr 18. PMID 22516508
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Efficacy (EFF) population is defined as all subjects in the Intent to Treat (ITT) population who enter into the Previous Antiepileptic (AED) Discontinuation (D/C) Phase. The Per Protocol (PP) population consists of all subjects in the EFF population who have no important protocol deviations related to efficacy.
Pre-assignment Details: Subjects are to be randomized into treatment with either Keppra XR 2000 mg/day or Keppra XR 1000 mg/day in a 3:1 ratio.
Groups:
- Keppra XR 1000 mg/Day: 1000 mg/day once daily for 18 weeks (administered as two Keppra XR tablets and two placebo tablets once daily)
- Keppra XR 2000 mg/Day: 2000 mg/day once daily for 18 weeks (administered as four Keppra XR tablets once daily)
Period: Overall Study
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Started | 57 (Number started refers to number randomized; 303 subjects were screened/enrolled and 228 randomized.) | 171
Completed | 50 | 141
Not Completed | 7 | 30
Not completed — Adverse Event | 3 | 7
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 14
Not completed — Withdrawal of consent | 1 | 5
Not completed — Other: Error determining exit criteria | 1 | 0
Not completed — Other: Patient non-compliant | 0 | 1
Not completed — Other: No contact for extended period | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day | Total
Number analyzed (Participants) | 57 | 171 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 31 | 42
  Between 18 and 65 years | 43 | 140 | 183
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.48 (16.32) | 34.31 (13.69) | 34.11 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 99 | 132
  Male | 24 | 72 | 96
Region of Enrollment [Number; unit: participants]
  United States | 8 | 29 | 37
  Mexico | 17 | 43 | 60
  Poland | 16 | 51 | 67
  Russian Federation | 16 | 48 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Exit Rate at 112 Days After the Beginning of the Previous Antiepileptic Drug (AED) Tapering Phase
Description: Cumulative exit rate at day 112, based on the duration between start date of previous AED tapering to the earliest date exit criterion was met; calculated using Kaplan Meier Methods. Subjects prematurely discontinued for reasons unrelated to exit criteria were censored as of last dose of study drug. Subjects who completed without meeting exit criteria were censored at Day 112. Exit criteria include increase in seizure frequency, severity, duration, status epilepticus, or new generalized seizure. Upper 95% 2-sided confidence limit for exit rate is compared to the historical control rate: 0.678.
Time Frame: 112 days
Population: Of the 171 (Keppra 2000 mg) subjects randomized, 158 subjects entered the Previous Antiepileptic Drug Tapering Phase and were included in the Efficacy Population. Primary Efficacy analysis was conducted for the Keppra XR 2000 mg/day group only.
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Number analyzed (Participants) | 0 | 158
proportion of subjects |  | 0.375 [0.297 to 0.453]

2. Secondary Outcome: The Cumulative Rate of Exit Events, Which Include Discontinuation Due to Exit Criteria, Withdrawal Due to Adverse Events (AE) and Withdrawal Due to Lack of Efficacy, at 112 Days After the Beginning of Previous Antiepileptic Drug (AED) Tapering Phase
Description: The cumulative exit event rate at Day 112 was calculated using Kaplan Meier methods. The exit event rate estimate was based on the duration between the start date of previous AED tapering to the earliest date an exit event occured. Subjects who prematurely discontinued for reasons unrelated to exit criteria, adverse event, or lack of efficacy were censored as of the last dose of study medication. Subjects who completed the study without having an exit event were censored as of Day 112.
Time Frame: 112 days
Population: Of the 171 (Keppra 2000 mg) subjects randomized, 158 subjects entered the Previous Antiepileptic Drug Tapering Phase and were included in the Efficacy Population. Evaluated for Keppra XR 2000 mg/day only.
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Number analyzed (Participants) | 0 | 158
proportion of subjects |  | 0.385 [0.307 to 0.463]

3. Secondary Outcome: The Cumulative Rate of Exit Events Due to Any Reasons at 112 Days After the Beginning of Previous Antiepileptic Drug (AED) Tapering Phase
Description: The cumulative exit event rate at Day 112 was calculated using Kaplan Meier methods. The exit event rate estimate was based on the duration between the start date of previous AED tapering to the earliest date an exit event occured. Subjects who completed the study without having an exit event were censored as of Day 112.
Time Frame: 112 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Number analyzed (Participants) | 0 | 158
proportion of subjects |  | 0.475 [0.397 to 0.553]

4. Secondary Outcome: The Cumulative Exit Rate at 112 Days for the Keppra XR 1000 mg Group After the Beginning of the Previous Antiepileptic Drug (AED) Tapering Phase
Description: Keppra XR 1000 mg arm was not intended for inferential analysis (planned 3 to 1 randomization, Keppra XR 2000 mg: 1000 mg). The Exit Rate was based on the duration between the start date of previous AED tapering to the earliest date an exit crterion was met. Subjects who prematurely discontinued for reasons unrelated to exit criteria were censored as of the last dose of study medication. Subjects who completed the study without meeting an exit criterion were censored as of Day 112.
Time Frame: 112 days
Population: Of the 57 (Keppra 1000 mg) subjects randomized, 54 subjects entered the Previous Antiepileptic Drug Tapering Phase and were included in the Efficacy Population.
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Number analyzed (Participants) | 54 | 0
proportion of subjects | 0.334 [0.204 to 0.465] |

ADVERSE EVENTS:
Time Frame: Up to 29 weeks
Arm/Group | Keppra XR 1000 mg/Day | Keppra XR 2000 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/57 | 12/171
Other Adverse Events (participants affected / at risk) | 33/57 | 87/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra XR 1000 mg/Day (N=57) | Keppra XR 2000 mg/Day (N=171)
haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
convulsion (Nervous system disorders) | 1 (1) | 4 (4)
status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra XR 1000 mg/Day (N=57) | Keppra XR 2000 mg/Day (N=171)
vertigo (Ear and labyrinth disorders) | 3 (3) | 7 (7)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (6)
irritablility (General disorders) | 3 (3) | 12 (12)
nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7)
somnolence (Nervous system disorders) | 12 (13) | 38 (40)
headache (Nervous system disorders) | 13 (34) | 32 (55)
convulsion (Nervous system disorders) | 9 (9) | 20 (20)
dizziness (Nervous system disorders) | 3 (4) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.